CLINICAL TRIAL: NCT04591002
Title: A Phase II, Study of Osimertinib to Suppress the Progression of Remaining Ground-glass Opacity Nodule (GGN) in Other Lobes After Curative Resection for Actionable EGFR Mutation-positive Stage IB-IIIA Lung Adenocarcinoma
Brief Title: Osimertinib to Suppress the Progression of GGN(EGFR Mutation-positive)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-19-20085
Record Dates: First submitted 2020-09-08; First posted 2020-10-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Osemertinib (Active Comparator)
  Interventions: Drug: Osimertinib 80 MG
- Observation (No Intervention)

INTERVENTIONS:
Drug: Osimertinib 80 MG — Osimertinib is an oral, potent, selective, irreversible inhibitor of both EGFR-TKI sensitising and resistance mutations in NSCLC with a significant selectivity margin over wild-type EGFR. Osimertinib will be administered orally as one 80 mg tablet once a day (1 cycle is 28 days). Cycles are repeated until disease progression, unacceptable toxicity, or until 1 year after the initiation of osimertinib administration.
  Arms: Osemertinib

SUMMARY:
This study designed to assess the efficacy of osimertinib (80 mg, orally, once daily) to suppress the progression of remaining GGN(s) in other lobes following surgical resection for actionable EGFR mutation-positive stage I lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Adult male or female patients, aged from 30 to 75 years
3. Pathologic proven stage I lung adenocarcinoma with additional persistent GGNs in at least one other lobe: GGN is defined as a ground glass-opacity with well-defined margin, mean density above -500 HU and greater than 7.5 mm in its maximum diameter
4. The resected lung adenocarcinoma should have actionable EGFR mutation, which is limited to L858R or exon 19 deletion.
5. WHO performance status 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks
6. Uneventful recovery from curative-intent lung cancer surgery
7. Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of childbearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation Further information in Appendix E (Definition of Women of Childbearing Potential and Acceptable Contraceptive Methods)
8. Male subjects should be willing to use barrier contraception (see Restrictions, Section 3.8)

Exclusion Criteria:

1. Treatment with any neoadjuvant therapy (radiation, any cytotoxic chemotherapy, investigational agents or other anticancer drugs after surgery) before randomization
2. Treatment with any adjuvant therapy (any cytotoxic chemotherapy, investigational agents or other anticancer drugs after surgery) before randomization
3. Extensive surgery other than lobectomy or sublobar resection (i.e. bilobectomy, sleeve lobectomy, pneumonectomy)
4. Past history of postoperative ALI/ARDS or pneumonia during recovery period
5. Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 week prior) (Appendix C). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foodswith known inducer effects on CYP3A4.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
8. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value. Whenever QTc, is mentioned in this document, this refers to correction e made by Fridericia formula (QTcF),
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
   * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN) , congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes
9. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
10. Inadequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count <1.5 x 109/L;
    * Platelet count <100 x 109/L;
    * Haemoglobin <90 g/L;
    * Alanine aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
    * Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
    * Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinaemia] or liver metastases;
    * Serum creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min [measured or calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
11. Women who are breast-feeding.
12. Males and females of reproductive potential who are not using and effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry.
13. Involvement in the planning and conduct of the study (applies to AstraZeneca staff or staff at the study site).
14. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of osimertinib on the regression of additional GGN(s) | up to 12months
  Regression rate of additional GGNs using investigator assessments by comparing the size of GGN(s) on the initial CT scan (at randomization) to that in the last follow-up scan. We will conduct the quantitative analysis of GGNs on the initial and follow-up CT scans via VOI (Volume of Interest) segmentation. VOI is measured with the unit of mm3.

SECONDARY OUTCOMES:
To assess the efficacy of osimertinib in avoidance of subsequent anticancer treatments including surgery or radiation for GGN(s) | up to 12months
  Avoidance rate of subsequent surgeries or radiation treatments for GGN(s) within one year since the initiation of osimertinib treatment: Defined as the number (percent) of patients who do not require subsequent anticancer treatments including surgeries or radiation for remaining GGN(s) within one year since the initiation of osimertinib treatment
To evaluate when GGN(s) will regress after osimertinib treatment | up to 12months
  Time to regression: Defined as the length of time from the date of initiation of osimertinib treatment to the first date of GGN regression
To evaluate the rate of treatment failure | up to 12months
  Incidence of regrowth and reappearance of remaining GGN(s) within one year since the initiation of osimertinib treatment
To evaluate the number of patients with new nodules | up to 12months
  Number of patients who would have growing new nodules (either ground glass nodules or solid nodules) with high suggestion of lung cancer by lung-special radiologists within one year since the initiation of Osimertinib treatment
To assess the incidence of treatment-emergent adverse events of osimertinib | up to 12months
  Incidence of adverse events and grades based on CTCAE (Common Terminology Criteria for Adverse Events) version 5.0.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - SMC, Seoul, Kangnamgu
  - Samsung medical center, Seoul

IPD SHARING:
Plan to Share IPD: No